CLINICAL TRIAL: NCT02801461
Title: The Effect of Extracorporeal Shock Wave Therapy in Patients With Cubital Tunnel Syndrome
Brief Title: The Effect of ESWT for Cubital Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending physician of physical medicine and rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 2-105-05-032
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Three-sessions of ESWT (Experimental): ESWT was given once a week for 3 weeks.
  Interventions: Device: extracorporeal shock wave therapy
- One-session of ESWT (Active Comparator): Single ESWT was given.
  Interventions: Device: extracorporeal shock wave therapy

INTERVENTIONS:
Device: extracorporeal shock wave therapy — Shock waves are defined a sequence of acoustic pulse characterized by a high peak pressure (100 MPa), fast pressure rise (< 10 ns) and short duration (10 μs).

SUMMARY:
The shock wave is a new and potential intervention for the reinnervation of peripheral nerve. The purpose of this study was to assess the effect of extracorporeal shock wave therapy on cubital tunnel syndrome.

DETAILED DESCRIPTION:
Investigators perform a prospective randomized, single-blinded study to investigate the effect of ESWT in patients with cubital tunnel syndrome.

Patients were randomized into intervention and control group. Participants in intervention group received three-sessions of ESWT and single one session of ESWT was given in control group. The evaluation was performed pretreatment as well as on the 4th, 8th, 12th, 16th and 24 week after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-80 year-old.
2. Typical symptoms and signs of cubital tunnel, such as positive Tinel's sign numbness/tingling in at least 5th digits, and in whom the diagnosis was confirmed using an electrophysiological study.

Exclusion Criteria:

1. Cancer
2. Coagulopathy
3. Pregnancy
4. Inflammation status
5. Patients who had conditions mimicking cubital tunnel syndrome, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome or who had previously undergone wrist surgery or steroid injection for cubital tunnel syndrome.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 4th, 8th, 12th, 16th and 24th weeks after treatment | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Visual analog scale (VAS)

SECONDARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  Using the Disabilities of the Arm, Shoulder and Hand to measure the symptoms and functional status before treatment and multiple time frame after treatment.
Change from baseline of electrophysiological study on 4th, 8th, 12th, 16th and 24th weeks | Pre-treatment, 4th, 8th, 12th, 16th and 24th weeks after treatment
  electrophysiological study according to the protocol reported by the American Academy of Neurology with SierraWave, Cadwell (USA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu YT, Ke MJ, Chou YC, Chang CY, Lin CY, Li TY, Shih FM, Chen LC. Effect of radial shock wave therapy for carpal tunnel syndrome: A prospective randomized, double-blind, placebo-controlled trial. J Orthop Res. 2016 Jun;34(6):977-84. doi: 10.1002/jor.23113. Epub 2015 Dec 10. PMID 26610183
- [Background] Assmus H, Antoniadis G, Bischoff C, Hoffmann R, Martini AK, Preissler P, Scheglmann K, Schwerdtfeger K, Wessels KD, Wustner-Hofmann M. Cubital tunnel syndrome - a review and management guidelines. Cent Eur Neurosurg. 2011 May;72(2):90-8. doi: 10.1055/s-0031-1271800. Epub 2011 May 4. PMID 21547883